CLINICAL TRIAL: NCT01107431
Title: A Combination of L-Arabinose and Chromium Lowers Circulating Glucose and Insulin Levels After Acute Oral Sucrose Challenge
Brief Title: Effects of a Dietary Supplement Containing L-Arabinose and Trivalent Patented Food-source of Chromium on Blood Glucose and Insulin
Acronym: L-Arabinose
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrative Health Technologies, Inc. (Network)
Responsible Party: Gilbert R. Kaats, PhD, Integrative Health Technologies, Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pharmachem 40-47
Record Dates: First submitted 2010-04-19; First posted 2010-04-21 (Estimated); Last update posted 2011-05-13 (Estimated); Status verified 2011-05

CONDITIONS: Pre-diabetes
Keywords: glucose; insulin; L-arabinose; Chromium
MeSH Terms: conditions — Glucose Intolerance; Insulin Resistance | interventions — Arabinose; Chromium; Sucrose; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sucrose with Dietary Supplement (Active Comparator): Repeated measures on subjects taking 70 grams of sucrose along with taking a dietary supplement containing L-Arabinose and Chromium
  Interventions: Dietary Supplement: L-Arabinose and Chromium
- Sucrose without Dietary Supplement (Active Comparator): Consumed 70 grams of sucrose without simultaneously taking the dietary supplement
  Interventions: Dietary Supplement: Sucrose without dietary Supplement

INTERVENTIONS:
Dietary Supplement: L-Arabinose and Chromium — Consumed 70 grams of sucrose simultaneously taking a dietary supplement
  Other Names: 70 grams of cane sugar along with supplement
  Arms: Sucrose with Dietary Supplement
Dietary Supplement: Sucrose without dietary Supplement — Repeated measures on subjects taking 70 grams of sucrose along with taking a dietary supplement containing L-Arabinose and Chromium
  Other Names: 70 grams of cane sugar with supplement
  Arms: Sucrose without Dietary Supplement

SUMMARY:
This study was designed to examine changes in capillary blood glucose and venous insulin levels after a 70 gram oral sucrose challenge with and without simultaneous consumption of a dietary supplement containing L-Arabinose and a patented version of chromium (LA-Cr).

DETAILED DESCRIPTION:
This study concluded that consumption of the LA-Cr supplement in conjunction with a 70-gram sucrose challenge led to a significant reduction of capillary blood glucose and venous insulin as compared to the sucrose challenge without the LA-Cr supplement. This finding may provide an important tool to reduce the adverse effects associated with elevated glucose and insulin levels.

ELIGIBILITY:
Inclusion Criteria:

* All study subjects were required to contact their family physician to ensure they had no medical conditions that would preclude their participation.

Exclusion Criteria:

* Diabetics, and
* Those not approved by their physicians.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2008-12; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Fasting Blood Glucose | Every 15 to 30 minutes
  Finger-stick glucose measurements taken every 15 or 30 minutes after taking a 70 gram sucrose challenge with and without the dietary supplement

SECONDARY OUTCOMES:
Fasting Blood Insulin Levels | Every 30 minutes
  A venipuncture blood test taken 30, 60, 90 and 120 minutes after taking a 70 gram sucrose challenge with and without taking the dietary supplement

CONTACTS AND LOCATIONS:
Overall Officials: Gilbert R Kaats, PhD, Principal Investigator — Integrative Health Technologies; Harry G Preuss, MD, Principal Investigator — Georgetown University
Locations (1):
- Integrative Health Technologies, San Antonio, Texas, United States

REFERENCES:
- [Derived] Kaats GR, Keith SC, Keith PL, Leckie RB, Perricone NV, Preuss HG. A combination of l-arabinose and chromium lowers circulating glucose and insulin levels after an acute oral sucrose challenge. Nutr J. 2011 May 6;10:42. doi: 10.1186/1475-2891-10-42. PMID 21548959